CLINICAL TRIAL: NCT02988245
Title: Prospective Randomized Controlled Trial Investigating the Use of Genetic Predisposition to Guide Pharmacologic Therapy for Hypertension
Brief Title: Investigating the Use of Genetics to Guide Pharmacologic Therapy for Hypertension
Acronym: PGEN for HTN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Geneticure, LLC (Industry)
Collaborators: Fairview Health Services (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Geneticure
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genetically-Guided Treatment for HTN (Experimental): Using a patient's genetic composition to guide BP prescribing for patients with hypertension, post diagnosis.
  Interventions: Drug: Geneticure Panel for HTN therapy
- JNC-8-Guided Treatment (Active Comparator): Using traditional (JNC-8) guidelines for BP prescribing for patients with hypertension, post diagnosis.
  Interventions: Drug: JNC-8

INTERVENTIONS:
Drug: Geneticure Panel for HTN therapy — Using either Genetics (Geneticure for HTN multi-gene panel) or JNC-8 guidelines for prescribing for patients with hypertension
  Arms: Genetically-Guided Treatment for HTN
Drug: JNC-8 — Using JNC-8 guidelines to guide therapy
  Arms: JNC-8-Guided Treatment

SUMMARY:
Hypertension is one of the most important preventable contributors to disease and death in the United States and represents the most common condition seen in the primary care setting. Approximately 78 million adults living in the U.S. have hypertension with more than 5 million new diagnoses made each year. Unfortunately, despite a significant impulse in the medical community to move towards an "individualized medicine" approach to patient centered treatment, the current clinical treatment strategy is based on a set algorithm which does not take into account individual patient differences. As a result hypertension is often sub-optimally treated based on "population averages", rather than a person's genetic make-up, with significant burden on our health care system. In fact, 40% of patients who are adherent to their blood pressure therapy (taking their medicines as prescribed by their clinician) do not have their blood pressure under control. Previous work has demonstrated significant functional polymorphisms within the kidney, vessels, and heart that will likely predict a patient's response to blood pressure pharmacotherapy. Previous work by our group, utilizing a retrospective design, has determined that the addition of genetic knowledge to prescribing can improve therapeutic guidance and decrease the time to blood pressure control significantly. Despite this, to date, there are no prospective trials to guide blood pressure therapy using multiple organ systems that are important in the three most common classes of drugs: diuretics, vasodilators, and beta-blockers. The objective of this clinical trial is to determine the efficacy of genetically guided therapeutic options for pharmacologic treatment of essential hypertension in newly diagnosed patients.

DETAILED DESCRIPTION:
Specific Aim:

To determine the efficacy of genetically guided therapeutic options for pharmacologic treatment of essential hypertension, when compared to conventional standard of care (JNC 8 guideline directed therapy).

Hypothesis A: Patients randomized to genetically guided blood pressure therapy will have significantly reduced time to optimal blood pressure control compared to conventional standard of care.

Hypotheses B: Patients randomized to genetically guided blood pressure therapy will have significantly greater absolute blood pressure reduction compared to conventional standard of care.

Hypothesis C: Patients randomized to genetically guided blood pressure therapy will have to take fewer classes of blood pressure medicines in order to achieve blood pressure control.

Secondary Aim:

To determine if genetically guided blood pressure therapy reduces number of medication changes in patients with hypertension.

Hypotheses: Patients randomized to genetically guided blood pressure therapy will have significantly less medication changes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with new diagnosis of hypertension or uncontrolled hypertension and on one medication
2. Subject is able and willing to provide informed consent
3. Subject is ≥ 30 and ≤ 80 years of age
4. Subject with a Body Mass Index (BMI) ≥ 19 and ≤ 50

Exclusion Criteria:

1. Subject has been diagnosed with chronic kidney disease as determined by serum creatinine levels of >1.3 mg/dl for men and >1.1 for women.
2. Subject has clinically significant cardiac disease as determined by diagnosed coronary artery disease, diagnosed heart failure, and congenital cardiac disease.
3. Subject has clinically significant vascular disease as determined by diagnosed peripheral vascular disease and diagnosed pulmonary hypertension.
4. Liver dysfunction is defined using the normal reference range for lower limit of normal and upper limit of normal used by Fairview labs and as determined by diagnosed liver disease /cirrhosis as listed in the patient's problem list based on ICD-10.
5. Subject has secondary hypertension.
6. Subject has prior diagnosis of endocrine disorders except uncomplicated type 2 diabetes and well controlled hypothyroidism.
7. Subject is pregnant.
8. Subject is breastfeeding.
9. Subject becomes pregnant during study
10. Subjects lacking the capacity to consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time to Blood Pressure Control | 1 year
  Time to BP control between genetically-guided prescribing and JNC-8 guided prescribing
Change in Blood Pressure | 1 year
  Change (absolute) in BP (systolic, SBP, diastolic, DBP, and mean arterial, MAP) between genetically-guided prescribing and JNC-8 guided prescribing
Number of Blood Pressure Medicines | 1 year
  Number of blood pressure medicines needed to obtain control of hypertension between genetically-guided prescribing and JNC-8 guided prescribing

SECONDARY OUTCOMES:
Number of Medication Changes | 1 year
  Number of blood pressure medicine changes needed to obtain control of hypertension between genetically-guided prescribing and JNC-8 guided prescribing

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Phelps, PharmD, Principal Investigator — Fairview Health Services; Weihong Tang, MD, PhD, Study Director — University of Minnesota; Michael Schulenberg, MD, Principal Investigator — Fairview Health Services
Locations (15):
- United States (15):
  - Fairview Health Clinics - Andover, Andover, Minnesota
  - Fairview Health Clinics - Blaine, Blaine, Minnesota
  - Fairview Health Clinics - Bloomington, Oxboro, Bloomington, Minnesota
  - Fairview Clinics - Brooklyn Park, Brooklyn Park, Minnesota
  - Fairview Clinics- Burnsville, Burnsville, Minnesota
  - Fairview Clinics - Columbia Heights, Columbia Heights, Minnesota
  - Fairview Health Clinics - Edina, Edina, Minnesota
  - Fairview Health Clinics - Elk River, Elk River, Minnesota
  - Fairview Clinics - Fridley, Fridley, Minnesota
  - Fairview Clinics - Lino Lakes, Lino Lakes, Minnesota
  - Fairview Clinics - Hiawatha, Minneapolis, Minnesota
  - Fairview Clinic - New Brighton, New Brighton, Minnesota
  - Fairview Clinics - North Branch, North Branch, Minnesota
  - Fairview Clinics - Wyoming, Wyoming, Minnesota
  - Fairview Health Services - Zimmerman, Zimmerman, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Site — http://www.geneticure.com